CLINICAL TRIAL: NCT04636918
Title: Ikervis for Prophylaxis of Dry Eye Disease Due to Graft vs Host Disease Post Allogeneic Haemtopoietic Stem Cell Transplant
Brief Title: Ikervis for DED Due to GVHD Post Allo-HSCT
Acronym: Ikervis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, Lim Li, Senior Consultant, Department of Corneal & External Eye Disease, Refractive surgery, Cataract & Comprehensive Ophthalmology, Adj Clinical Investigator, Adj A/Professor, Singapore Eye Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R1641/38/2019
Record Dates: First submitted 2020-03-09; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Leukemia (Both ALL and AML); MDS-EB-1
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Other): Ikervis (cyclosporine 0.1%), emulsion, one drop into both eyes, once at night.
  Interventions: Drug: Cyclosporine Ophthalmic

INTERVENTIONS:
Drug: Cyclosporine Ophthalmic — Prospective interventional study (single arm)
  Other Names: Ikervis

SUMMARY:
Dry eye disease (DED) is a common sequelae of graft versus host disease (GVHD) after allogeneic hematopoietic stem cell transplantation (allo-HSCT). Since Ikervis is reported to be a safe and efficacious treatment of DED associated with chronic GVHD, our study would like to study the efficacy of prophlactic Ikervis in preventing ocular GVHD development.

DETAILED DESCRIPTION:
This is a prospective single arm interventional study.

The recruitment period will be over 12-18 months to enroll all suitable patients. The total duration of prophylaxis will be for 1 year. After completion of the period of prophylaxis, the patients will be followed up as a non-study patient as clinically indicated.

Forty subjects, undergoing allo-HSCT, will be recruited from the Singapore National Eye Centre upon referral from the Department of Hematology, Singapore General Hospital and followed up at least 5 times over a period of 12 months at the Singapore Eye Research Institute.

The images of the subject eyes will be recorded and stored electronically. These images (corneal fluorescein staining score, Lipiview, meibography, conjunctival redness, tear stability assessment) will be used in the analysis of outcome measures. The Lipiview result is in video format.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 and above
* Able to give informed consent

Exclusion Criteria:

* Presence of concurrent disease
* Unable to complete the follow up

Ages: 13 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2022-08-22 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess change in basline visual acuity using LogMAR chart with prophylactic Ikervis after 3 to 5 weeks before Haematopoietic Stem Cell Transplant and 3 months, 6 months and 12 months post Haematopoietic Stem Cell Transplant. | Baseline, 3 months, 6 months and 1 year post-HSCT follow up
  Visual acuity will be assessed using LogMAR chart at baseline screening and 3, 6, and 12 months post-HSCT after prophylactic Ikervis.
To assess change in baseline intraocular pressure using non-contact tonometry with 3 months, 6 months and 12 months post Haematopoietic Stem Cell Transplant. | Baseline, 3 months, 6 months and 1 year post-HSCT follow up
  Intraocular pressure (mmHg) will be assessed using non-contact tonometry at baseline screening and 3, 6, and 12 months post-HSCT after prophylactic Ikervis.
To assess change in baseline anterior ocular health using slit lamp examination with 12 months post Haematopoietic Stem Cell Transplant. | Baseline screening and 1 year post-HSCT follow up
  Slit lamp examination will be performed at baseline screening and 12 months post-HSCT after prophylactic Ikervis. Clinical findings such as macroerosions or chemosis on cornea, or cataract will be recorded.
To assess change in baseline posterior ocular health using fundus examination with 12 months post Haematopoietic Stem Cell Transplant. | Baseline screening and 1 year post-HSCT follow up
  Fundus examination will be performed at baseline screening and 12 months post-HSCT after prophylactic Ikervis. Clinical findings such as cup disc ratio will be graded from 0.0 to 1.0 (greater value means larger cup), hemorrhage, edema of the retina/macular will be recorded.
To assess change of baseline dry eye symptoms with prophylactic Ikervis after 3 to 5 weeks before Haematopoietic Stem Cell Transplant and 3 months, 6 months and 12 months post Haematopoietic Stem Cell Transplant. | Baseline, 3 to 5 weeks from baseline (Pre-HSCT), 3 months, 6 months and 1 year post-HSCT follow up
  Dry eye symptoms will be assessed using SPEED questionnaire (in score 0-28). A higher score means worse dry eye symptom. The change of dry eye symptoms will be assess from baseline before prophylactic Ikervis, 3 to 5 weeks from baseline (Pre-HSCT), and 3, 6, and 12 months post-HSCT after prophylactic Ikervis.
To assess change of baseline non-invasive tear break up time with prophylactic Ikervis after 3 to 5 weeks before Haematopoietic Stem Cell Transplant and 3 months, 6 months and 12 months post Haematopoietic Stem Cell Transplant. | Baseline, 3 to 5 weeks from baseline (Pre-HSCT), 3 months, 6 months and 1 year post-HSCT follow up
  Non-invasive tear break up time (in seconds) will be assessed using Oculus Keratography K5M. The change of NITBUT will be assessed from baseline before prophylactic Ikervis, pre-HSCT, and 3, 6, and 12 months post-HSCT after prophylactic Ikervis.
To assess change of baseline conjunctival redness with prophylactic Ikervis after 3 to 5 weeks before Haematopoietic Stem Cell Transplant and 3 months, 6 months and 12 months post Haematopoietic Stem Cell Transplant. | Baseline, 3 to 5 weeks from baseline (Pre-HSCT), 3 months, 6 months and 1 year post-HSCT follow up
  Conjunctival Redness (in grading 0-4) will be assessed using Oculus Keratography K5M. A higher grading means conjunctiva is more red. The change of conjunctival redness will be assessed from baseline before prophylactic Ikervis, pre-HSCT, and 3, 6, and 12 months post-HSCT after prophylactic Ikervis.
To assess change of baseline tear lipid thickness with prophylactic Ikervis 12 months post Haematopoietic Stem Cell Transplant. | Baseline and 1 year post-HSCT follow up
  Tear lipid thickness will be measured using LipiView. The change of tear lipid thickness will be only be assessed from baseline before prophylactic Ikervis and 12 months post-HSCT after prophylactic Ikervis.
To assess change of baseline Meibomian gland status with prophylactic Ikervis 12 months post Haematopoietic Stem Cell Transplant. | Baseline and 1 year post-HSCT follow up
  Meibomian gland (in grade 0-3) will be assessed using Infra-red Meibography. We will grade the Meibomian gland disease as: 0, no loss of meibomian glands; 1, lost area was less than one third of the total area of meibomian glands; 2, lost area was between one third and two thirds of the total area of meibomian glands; 3, lost area was over two thirds of the total area of meibomian glands. The change of meibomian gland will be assessed from baseline before prophylactic Ikervis pre-HSCT and 12 months post-HSCT after prophylactic Ikervis.
To assess change of baseline tear cytokines with prophylactic Ikervis after 3 to 5 weeks after 3 to 5 weeks before Haematopoietic Stem Cell Transplant and 3 months, 6 months and 12 months post Haematopoietic Stem Cell Transplant. | Baseline, 3 to 5 weeks from baseline (Pre-HSCT), 3 months, 6 months and 1 year post-HSCT follow up
  Tear cytokine will be analysed with tears extracted from Schirmers test. The change of tear cytokines will be assess from baseline before prophylactic Ikervis, 3 to 5 weeks from baseline (Pre-HSCT), and 3, 6, and 12 months post-HSCT after prophylactic Ikervis.
To assess change of conjunctival impression cytology 3 to 5 weeks after prophylactic Ikervis with 12 months post Haematopoietic Stem Cell Transplant. | 3 to 5 weeks from baseline (Pre-HSCT) and 1 year post-HSCT follow up
  Conjunctival impression cytology will be performed using EyePrim. The change of conjunctival impression cytology only will be assessed 3 to 5 weeks from baseline (Pre-HSCT) and 12 months post-HSCT after prophylactic Ikervis.
To assess change of baseline corneal fluorescein staining score with prophylactic Ikervis after 3 to 5 weeks before Haematopoietic Stem Cell Transplant and 3 months, 6 months and 12 months post Haematopoietic Stem Cell Transplant. | Baseline, 3 to 5 weeks from baseline (Pre-HSCT), 3 months, 6 months and 1 year post-HSCT follow up
  Corneal fluorescein staining (in grade 0-4) will be imaged by Oculus Keratograph K5M. A greater number indicating more intense or greater area of staining. The change of corneal fluorescein staining will be assess from baseline before prophylactic Ikervis, 3 to 5 weeks from baseline (Pre-HSCT), and 3, 6, and 12 months post-HSCT after prophylactic Ikervis.
To assess change of baseline Meibomian gland expressibility with prophylactic Ikervis after 3 to 5 weeks before Haematopoietic Stem Cell Transplant and 3 months, 6 months and 12 months post Haematopoietic Stem Cell Transplant. | Baseline, 3 to 5 weeks from baseline (Pre-HSCT), 3 months, 6 months and 1 year post-HSCT follow up
  Meibomian gland expressibility will be assessed using Meibomian gland evaluator. Texture of expressed secretion will be graded as liquid or viscous. The number of expressible glands will be recorded. The change of meibomian gland expressibility will be assess from baseline before prophylactic Ikervis, 3 to 5 weeks from baseline (Pre-HSCT), and 3, 6, and 12 months post-HSCT after prophylactic Ikervis.
To assess Quality of Life Questionnaire at 12 months post Haematopoietic Stem Cell Transplant. | 1 year post-HSCT follow up
  Quality of Life (in score 0, 1, 2, 3, 8) will be assessed using Impact of Vision Impairment Profile questionnaire at the end of the prophylactic Ikervis, 12 months post-HSCT. The score in 0 means a lot of the time, 1 means a fair amount of the time, 2 means a little of the time, 3 means not at all, 8 means do not do this for other reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Li Lim, Principal Investigator — Senior Consultant
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tong L, Lim EWL, Yeo SWJ, Hou A, Linn YC, Ho A, Than H, Quek JKS, Hwang WYK, Lim FLWI, Lim L. Conjunctival T Cell Profile in Allogeneic Hematopoietic Stem Cell Transplant Patients after Instilling Topical Cyclosporine-A 0.1% Cationic Emulsion. Ophthalmol Ther. 2023 Jun;12(3):1547-1567. doi: 10.1007/s40123-023-00686-0. Epub 2023 Mar 1. PMID 36856978